CLINICAL TRIAL: NCT05917080
Title: Efficacy of Neuromuscular Training and Manual Therapy With Augmented Low-Dye Taping Technique for Correction of Pronated Foot in the Management of Anterior Knee Pain
Acronym: AKPS NPRS FPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mediclinic Al Noor Hospital (Other)
Responsible Party: Principal Investigator, Albert Anand.U, Physiotherapy Team Lead - Principal Investigator, Mediclinic Al Noor Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCME.CR.310.MNOO.2023
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Anterior Knee Pain Syndrome; Pronated Foot
Keywords: Anterior Knee pain; Pronated foot; Manual therapy; Neuro muscular exercise; low dye taping; Foot Posture index; Numerical pain rating scale; dynamic Knee valgus angle; Kujala Scale
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Biomechanical Relationship of pronated foot & Anterior knee pain
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental Group) (Experimental): Manual Therapy Technique Anti-Pronation Low- Dye Taping Technique Intrinsic Foot Muscles Exercises Calf Muscle & Plantar Fascia Stretching VMO Strengthening
  Interventions: Other: Manual Therapy
- Group B (Experimental Group) (Experimental): Neuromuscular Training Anti-Pronation Low- Dye Taping Technique Intrinsic Foot Muscles Exercises Calf Muscle & Plantar Fascia Stretching VMO Strengthening
  Interventions: Other: Manual Therapy
- Group C (Control Group) (Other): Intrinsic Foot Muscles Exercises Calf Muscle & Plantar Fascia Stretching VMO Strengthening
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — Manual Therapy: Manual therapy is the use of hands-on techniques to evaluate, treat, and improve the status of Neuro-musculoskeletal conditions.
  Augmented Low-Dye Taping: Augmented Low-Dye taping is designed to off-load the plantar fascia & applied below the ankle and is hypothesised to generate a supinating force that controls the amount of pronation at the subtalar joint.
  Neuromuscular Exercises: Neuromuscular training could be defined as training enhancing unconscious motor responses by stimulating both afferent signals and central mechanisms responsible for dynamic joint control.
  Strengthening Exercises:The strengthening of the muscles promotes better overall functioning of the foot and thereby can help to take some of the tension out of the fascia.
  Stretching exercises:Static stretching is defined as passively stretching a given muscle-tendon unit by slowly placing it maximal position of stretch and sustaining it there for an extended period of time.
  Other Names: Neuromuscular Training Anti-Pronation Low- Dye Taping Technique Intrinsic Foot Muscles Exercises Calf Muscle & Plantar Fascia Stretching VMO Strengthening

SUMMARY:
The goal of this clinical trial] is to To find out the effect of Neuromuscular Training and Manual therapy with Augmented Low - Dye Taping technique for correction of Pronated foot in the management of Anterior knee pain patients. The main question[s] it aims to answer are:

* Is there any Kinematic association of biomechanical risk factors between anterior knee pain & pronated foot?
* Is there any potential impact of therapeutic foot interventions for correction of Pronated foot in the management of anterior knee pain?

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is one of the most prevalent musculoskeletal injuries seen by physiotherapists and sport medicine practitioners. The PFPS occurs in 17% of male and 33% of female knee pathology. The pain is usually aggravated by activities involving patellofemoral compressive forces such as remaining in the sitting position with the knees flexed for long periods of time (movie goers sign). Patellofemoral pain syndrome (PFPS) is an important clinical problem and the most prevalent disorder of the knee.

The etiology of PFPS is not fully understood and may consist of multiple factors including lower leg and foot malalignment. Patella femoral pain syndrome (PFPS) may arise from abnormal muscular and biomechanical factors that alter tracking of the patella within the femoral trochlear notch contributing to increased patellofemoral contact pressures that result in pain and dysfunction.

Excessive foot pronation during gait is frequently linked to patellofemoral pain syndrome (PFPS) development, due a proposed coupling of increased foot pronation with increased tibial and femoral internal rotation. This excessive pronation can result in increased soft tissue stress and changes in overall lower limb alignment, often predisposing the individual in question to injury of the lower extremity. Excessive rear foot pronation therefore may lead to abnormal tibia internal rotation which could possibly translate to greater stress on the knee structure, altering patella tracking. Excessive pronation of the subtalar joint particularly is thought to lead to patellofemoral disorders. The excessive subtalar joint pronation may delay external rotation of the leg, and therefore will inhibit supination of the foot. Physiotherapy consisted of a combined therapy approach that has proved efficacious in patellofemoral pain syndrome. Physical therapy is the mainstay in non-operative treatment.

Joint proprioceptors have historically been considered "limit detectors", stimulated at the extremes of joint range-of-motion (ROM). Joint proprioceptors provide input throughout a joint's entire ROM under both low and high load conditions stimulating strong discharges from the muscle spindle and are thus vital for joint stability.

The augmented low-Dye (ALD) is a taping technique frequently used by clinicians in the management of lower limb musculoskeletal pain and injury. A recent review of the literature concluded that ALD tape produces a biomechanical effect, specifically by increasing medial longitudinal arch height, reducing calcaneal eversion and tibial internal rotation, reducing medial forefoot pressures and increasing lateral midfoot pressures during standing, walking and jogging. The LD taping technique aims to reduce excessive pronation by creating an external supinating force medial to the subtalar joint axis, namely at the medial plantar surface of the foot.

Patients with plantar heel pain treated with the manual therapy demonstrated complete pain relief and full return to activities. Manual therapy helps in bringing back the malalignment of the foot and correcting foot problems which intern reduces the heel pain.

The Aim of the study is to find out the effect of Neuromuscular Training and Manual therapy with Augmented Low - Dye Taping technique for correction of Pronated foot in the management of Anterior knee pain. The previously available studies are mainly limited to foot orthoses & focused on the knee joint interventions. There is a lack of research related to therapeutic interventions for the foot, an intrinsic risk factor, can address the fundamental component of anterior knee pain.

The Novelty of Study is to the find out potential impact of therapeutic foot interventions for correction of Pronated foot in the management of anterior knee pain.

The Objectives of the study is followed below

* To find out the association of biomechanical risk factors between Anterior knee pain & pronated foot.
* To find out the effect of Manual therapy with Augmented Low- Dye taping technique on the selective outcome parameters.
* To find out the effect of Neuromuscular Training with Augmented Low- Dye taping technique on the selective outcome parameters.
* To compare the effect of Manual therapy and Neuromuscular Training with Augmented Low- Dye taping technique on the selective outcome parameters.

Null Hypothesis:

• There is no significant improvement in the pain and functional Limitations, following Manual therapy & Neuro muscular training with Augmented Low - Dye Taping technique for correction of Pronated foot in the management of Anterior knee pain.

Alternative Hypothesis:

• There is a significant improvement in the pain and functional Limitations, following Manual therapy & Neuro muscular training with Augmented Low - Dye Taping technique for correction of Pronated foot in the management of Anterior knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 to 35 years
* Sex - both males & females
* Clinically diagnosed patient of PFPS with Pronated foot
* Anterior or posterior pain in the knee area lasting for more than 12 weeks
* Excessive calcaneal eversion measured at 6° in the relaxed posture
* Score of between three and seven points on the numerical pain rating in activities of daily living Kujala Scale Point 40 & Above

Exclusion Criteria:

* A history of diagnosis of meniscus or joint injury & knee joint surgery
* Taking nonsteroidal anti-inflammatory drugs or corticosteroids within 24 hrs before the test
* History of brain injury or vestibular disorder within the last 6 months
* Positive sign of Patellar Apprehension test
* Congenital or traumatic deformity
* Allergic reactions to taping
* Concomitant diagnosis of pre patellar bursitis or tendonitis
* knee Ligamentous injury or laxity
* Plica syndrome & Osgood Schlatter's disease
* Malignancy & Skin Infection
* Pregnant woman or lactating women.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
AKPS (Kujala Scale) | 6 months
  Anterior knee pain scale - measuring Functional Limitations, The AKPS contains 13 items self reported questionnaires. The AKPS graded on Scale of "0 to 100" with 100 being the highest possible score. lower scores reflect the greater pain & disability.
FPI | 6 months
  Foot Posture index - Analyzing the Foot posture - The FPI-6 is a novel method of rating foot posture using set criteria and a simple scale, and is a quick, reliable diagnostic tool. neutral foot posture are graded as zero, while Pronated postures are given a positive value, the higher the value the more pronated. For a neutral foot the final FPI aggregate score should lie somewhere around zero.
NPRS | 6 months
  Numerical Pain rating Scale-Measuring the pain. The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
DVI | 6 months
  Dynamic Valgus Index -Measuring the Dynamic knee valgus angulation. Two dimensional motion analysis of lower extremity movement typically focuses on the knee frontal plane projection angle, which considers the position of the femur and the tibia. A measure that includes the pelvis may provide a more comprehensive and accurate indicator of lower extremity movement. Dynamic knee valgus two-dimensional angular measures. 1a. Hip frontal plane projection angle, calculated as 90 ° minus the angle (α) between the pelvis segment and the thigh segment. Knee frontal plane projection angle, calculated as 180 ° minus the angle (β) between the thigh segment and the shank segment. 1b. Example of individual demonstrating an observable dynamic knee valgus, resulting in increased hip and knee frontal plane projection angles and a larger dynamic valgus index.

CONTACTS AND LOCATIONS:
Locations (1):
- Mediclinic Al Noor Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided